CLINICAL TRIAL: NCT03681314
Title: Long-term Outcomes of Umbilical Cord Milking in Term and Late Preterm Neonates Who Are Depressed at Birth
Brief Title: Umbilical Cord Milking in Neonates Who Are Depressed at Birth-Developmental Follow Up (MIDAB-FU)
Acronym: MIDAB-FU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was not funded. The same study with few modifications in the trial was later funded by the NICHD. Now study started enrolling babies using new registration and identification IDs ( NCT03682042 and NCT03657394).
Sponsor: Nemours Children's Clinic (Other)
Collaborators: NPKSIMS, Nagpur, India (Unknown); Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Zubair Aghai, Professor of Pediatrics, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCM2018FU
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Birth Asphyxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Neurodevelopmental assessments will be done at 2 years of age (22-26 months) for subjects who were randomized to receive either immediate cord clamping or umbilical cord milking as part of the MIDAB trial.
Who Masked: Outcomes Assessor
Masking Description: Neurodevelopmental providers will be blinded to the randomization of the toddler during the examination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Active Comparator): At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 10-15 seconds.
  Interventions: Other: Umbilical Cord Milking
- Immediate Cord Clamping (No Intervention): The umbilical cord is clamped immediately after the delivery.

INTERVENTIONS:
Other: Umbilical Cord Milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 10-15 seconds.
  Arms: Umbilical Cord Milking

SUMMARY:
An extension of the MIDAB trial, the MIDAB-Follow-up trial will evaluate the neurodevelopmental outcomes at 22-26 months age of term/late preterm infants who were depressed at birth and received umbilical cord milking (UCM) or immediate cord clamping (ICC).

DETAILED DESCRIPTION:
The MIDAB-Follow-up trial will examine the difference in survival and neurodevelopmental impairment of infants who were depressed at birth and enrolled in MIDAB trial. The difference in survival and neurodevelopmental impairment in infants who received UCM and ICC will be assessed using standardized neurological and developmental assessment tools at 22-26 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in MIDAB trial

Exclusion Criteria:

* None

Ages: 3 Months to 26 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-06-16 (Estimated); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental Outcome at 2 Years of Age | 22-26 months
  Overall and Domain Scores - Ages and Stages, 3rd ed. Questionnaire

SECONDARY OUTCOMES:
Fidgety Movements at 3 months of age | 3-5 months
  Assessment of Fidgety Movements by Prechtl's method
Neurodevelopmental Outcome at 1 Year of Age | 10-14 months
  Developmental Activities Screening Inventory - Second Edition (DASI-II)
Autism Outcome | 22-26 months
  Modified Checklist for Autism in Toddlers (M-CHAT-R)

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Aghai, MD, Principal Investigator — Nemours Children's Clinic
Locations (3):
- India (3):
  - Daga Memorial Woman and Children Hospital, Nagpur, MS
  - Government Medical College and Hospital, Nagpur, MS
  - NKP Salve Institute of Medical Sciences and Lata Mangeshkar Hospital, Nagpur, MS

IPD SHARING:
Plan to Share IPD: Undecided